CLINICAL TRIAL: NCT06096818
Title: The Effectiveness of Kegel Exercises and Abdominal Exercises on Stress Urinary Incontinence Severity, Quality of Life, and Sleep Quality In Menopausal Women With Urinary Incontinence
Brief Title: Kegel and Abdominal Exercises on Urinary Incontinence Severity, Quality of Life, and Sleep Quality in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Meltem Kaydırak, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B.30.2.ODM.0.20/60-164
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence; Postmenopausal Symptoms; Sleep Quality
Keywords: Menopause; Female; Urinary incontinence; Kegel Exercise; Abdomen Exercise
MeSH Terms: conditions — Urinary Incontinence; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Type of Study: This study is a randomized controlled trial. The pre-test-post-test has be carried out with a pattern.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Women who meet the inclusion criteria were included in the sample using a simple random method. Before the research numbers were produced from random.org, envelopes of the same size and characteristics were created for each participant by someone other than the researcher (IU-C, Research Assistant B.Y), and numbers between 1 and 100 were written on them. Then, considering the data losses, numbers from 1 to 100 were generated from random.org. Single-column groups were created between 1 and 100 by the help of the Random Integer Generator at the Numbers title of the Random.org website. The numbers (1 or 2) were assigned to the groups (study and control) randomly by tossing a coin. Number 1 was assigned to the control group, and number 2 to the experimental group.
  Experimental Group: 35 women Control Group: 35 women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Kegel exercises and abdominal exercises (Experimental): Kegel exercises and abdominal exercises training has given to this group
  Interventions: Behavioral: Experimental Group: Kegel exercises and abdominal exercises; Behavioral: Control Group: Kegel exercises
- Control Group: Kegel exercises (No Intervention): Kegel exercises exercises training has given to this group

INTERVENTIONS:
Behavioral: Experimental Group: Kegel exercises and abdominal exercises — The training was planned to occur 3 times in a 12-week period (first meeting+6thweek+12th week). Each training: approx. 30 min.
  First session:Meeting the woman Consent and data collection forms (Descriptive characteristics of women, Incontinence Impact Questionnaire-Short Form,International Urinary Incontinence Consultation Questionnaire-Short Form,Pittsburgh Sleep Quality Scale) Information about stress urinary incontinence is given The woman is given kegel exercise and abdominal exercise training face to face by the researchers.
  Kegel and abdominal exercise application chart is explained and given as homework.
  Relevant brochure is provided. Second Session:Greeting-Kegel and abdominal exercise application chart is being checked Kegel and abdominal exercises are performed again under the supervision of the researcher.
  Third session:Greeting-Kegel and abdominal exercise application chart is being checked Data collection tools are being refilled.
  Arms: Experimental Group: Kegel exercises and abdominal exercises
Behavioral: Control Group: Kegel exercises — The training was planned to occur 3 times in a 12-week period (first meeting+6th week+12th week). Each training: approx. 20 min.
  First session: Meeting the woman Consent and data collection forms (Descriptive characteristics of women, Incontinence Impact Questionnaire-Short Form, International Urinary Incontinence Consultation Questionnaire-Short Form, Pittsburgh Sleep Quality Scale).
  Information about stress urinary incontinence is given The woman is given kegel exercise training face to face by the researchers. Kegel exercise application chart is explained and given as homework. Relevant brochure is provided. Second Session:Greeting-Kegel exercise application chart is being checked Kegel exercises are performed again under the supervision of the researcher. Third session:Greeting-Kegel exercise application chart is being checked Data collection tools are being refilled.
  Arms: Experimental Group: Kegel exercises and abdominal exercises

SUMMARY:
The aim of this randomized, controlled experimental study is to investigate the effectiveness of Kegel exercises and abdominal exercises on urinary incontinence severity, quality of life, and sleep quality in menopausal women with stress urinary incontinence. Research Hypothesis are:

H1: Combining Kegel exercises and abdominal exercises affects urinary incontinence severity in menopausal women with stress urinary incontinence.

H2: Combining kegel exercises and abdominal exercises affects quality of life in menopausal women with stress urinary incontinence.

H3: Combining kegel exercises and abdominal exercises affects sleep quality in menopausal women with stress urinary incontinence.

Researchers will compare two groups: Kegel and abdominal exercise training is applied to the experimental group. Only kegel exercise training is applied to the control group.

The study will be conducted in a prospective, randomized, parallel group controlled design. Hypotheses will be evaluated by applying pre-test and post-tests to the groups of exercises applied for three months during the research process.

DETAILED DESCRIPTION:
Urinary incontinence is defined by the International Continence Society as involuntary urinary leakage that causes social and hygienic problems and can be objectively demonstrated. Urinary incontinence is an important health problem that is more common in women than men. As a matter of fact, urinary incontinence has also been recognized as a common public health problem affecting women's physical, psychological, social, and economic well-being. This problem may worsen, especially during menopause, as estrogen levels decrease and pelvic floor muscles and ligaments atrophy.

Women spend a long period of their lives in menopause. Therefore, the urinary incontinence they experience during this period affects their lives in many dimensions (insecurity, deterioration in sexual life, insomnia, etc.). As a matter of fact, one of the important conservative treatments for urinary incontinence is Kegel exercises. The fact that it has no risks or costs and that women can do it wherever and whenever they want makes this exercise advantageous. It has been reported that abdominal muscle exercises (bridge building and abdominal curling exercises, etc.), along with Kegel exercises, significantly affect the pelvic floor muscles. However, the studies are mostly on the samples of pregnant, postpartum, and reproductive-age women, and studies on women in the menopausal period are needed. This study will increase awareness of the importance and effect of regular kegel and abdominal exercises in menopausal women with urinary incontinence.

Deterioration in sleep quality and chronic insomnia are also quite common (11.8% - 56.6%) problems in menopause. One of the factors that cause sleep problems is urinary incontinence, which causes frequent trips to the toilet and interrupts night sleep. Researchers predicted that reducing the frequency of urinary incontinence experienced by women would positively affect their sleep quality.

Data Collection: The data will be collected by the researcher by face-to-face interview method in a total of 12 weeks, three face-to-face interviews, each interview is experimental group 30 minutes - the control group 20 minutes. Kegel and abdominal exercise training is applied to the experimental group. Only kegel exercise training is applied to the control group.

Statistical Methods to be Used: The Statistical Package for the Social Sciences program will be used to analyze the obtained data. The conformity of the data to the normal distribution will be examined by considering the Shapiro-Wilk test. Parametric methods will be used to analyze normally distributed variables, and non-parametric methods will be used to analyze non-normally distributed variables. Independent-sample T-test, Mann-Whitney U (Exact) test, and T-test for Dependent Groups, Wilcoxon test will be used to compare two independent groups. Pearson correlation Spearman's tests will be used to examine the correlations of the variables with each other. Comparison of categorical data will be tested with Pearson Chi-square and FisherExact tests.

ELIGIBILITY:
Criteria for inclusion in the study:

* Able to read and write,
* Without hearing difficulty or vision loss, Able to communicate,
* Those who have not received any treatment for incontinence,
* Having a body mass index (BMI) < 30,
* Those who have stage 0-I-II stress urinary incontinence complaints, who have been diagnosed with stress incontinence by a physician and who do not require surgical treatment for stress incontinence,
* Women in menopause who agree to participate in the study will be included in the study.

Criteria for exclusion from the study:

* Having diabetes,
* Those who use diuretics and antihypertensive drugs,
* Having a urinary system infection,
* Those with pelvic organ prolapse,
* Having undergone incontinence surgery,
* Those with lumbar disc herniation,
* Body mass index (BMI) > 30,
* Those who have stage III-IV stress urinary incontinence complaints, have been diagnosed and require surgical treatment for stress incontinence
* Women who do not agree to participate in the study and who are not in menopause will not be included in the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence Severity | The change in the International Consultation on Incontinence Questionnaire-Short Form score of the participants in 3 months was evaluated.
  70 women as assessed by International Consultation on Incontinence Questionnaire-Short Form, Change From Baseline in Urinary Incontinence Severity at 3 months. In menopausal women with urinary incontinence, performing kegel exercises and abdominal exercises together reduces the total score of the International Consultation on Incontinence Questionnaire-Short Form.
  The International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) consisting of 6 questions was used to assess the severity, frequency, type of incontinence and its implications on quality of life. The possible scores on the scale are between 0 and 21.
Quality of life of women with urinary incontinence will be evaluated | The change in the incontinence Impact Questionnaire-IIQ-7 score of the participants in 3 months was evaluated. Participants were expected to have an decrease in their scores during this time
  Incontinence Impact Questionnaire (IIQ-7): This scale is reliable, consistent and valid instrument to measure of the impact of urinary incontinence, to assess the impact on quality of life in Turkish speaking women with urinary incontinence. The Likert-type scale has four dimensions: physical activity, travel, social relations and emotional health. A minimum of 0 and a maximum of 21 points can be obtained from IIQ-7. The total score and sub-dimension scores of the form are calculated on a scale of 0 - 100 points. Low scores obtained from each IIQ-7 are an indicator of increased quality of life.
Sleep Quality | The change in the participants' sleep quality at 3 months was evaluated with The Pittsburgh Sleep Quality Scale. Participants were expected to have an decrease in their scores during this time.
  Pittsburgh Sleep Quality Scale (PSQI): It is a scale to evaluate sleep quality with questions asked under seven main headings that evaluate subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping pills and impairment in daytime functions. The total score of the scale is between 0-21. If the total score is 5 or above, sleep quality is considered poor. High scores indicate poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpaşa, Istanbul, Marmara Region, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The information obtained from this study will be used for research purposes and personal information will be kept confidential; however, the data may be used for publication purposes. 2 years after the completion of the study, the data will be destroyed by the destruction machine belonging to the institution and will be kept locked in a closed cabinet during this period.